CLINICAL TRIAL: NCT05507892
Title: Molecular Mechanisms of SGLT2 Inhibition in Diabetic Kidney Disease
Brief Title: Renal Mechanism of SGLT2 Inhibition
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-0668
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — Canagliflozin; p-Aminohippuric Acid

STUDY DESIGN:
Intervention Model Description: This is an open-label non-randomized mechanistic trial. This trial will enroll 40 participants who will receive 100 mg of canagliflozin daily for six (6) months in addition to standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants who will receive 100 mg of canagliflozin daily for six (6) months in addition to standard of care.
  Interventions: Drug: canagliflozin; Drug: Aminohippurate Sodium Inj 20%

INTERVENTIONS:
Drug: canagliflozin — Canagliflozin is in a class of medications called sodium-glucose co-transporter 2 (SGLT2) inhibitors. It is a used to treat type 2 diabetes. Canagliflozin lowers blood sugars by causing the kidneys to excrete more glucose in the urine.
  Other Names: Invokana
Drug: Aminohippurate Sodium Inj 20% — Diagnostic aid/agent used to measure renal plasma flow (RPF) PAH (Basic Pharma, Geleen, Netherlands) has been used to measure RPF in human research for 7 decades, and is very well tolerated and generally recognized as safe with low toxicity.
  Other Names: -Sodium 4-amino hippurate (PAH) inj 20% 2g/10mL -Para-aminohippurate

SUMMARY:
Canagliflozin is an oral drug which is currently approved for use in patients with type 2 diabetes by the US Food and Drug Administration (FDA). Canagliflozin acts by increasing salt and sugar loss in the urine, and has shown to protect heart, kidney, and blood vessel function in patients with type 2 diabetes. However, it is unknown how canagliflozin protects the kidneys from disease. Therefore, this study plans to learn more about how canagliflozin works to protect against diabetic kidney disease in adults with type 2 diabetes. This study will use state-of-the-art kidney imaging, kidney biopsies and detailed testing of kidney function to determine the mechanisms of protection afforded by canagliflozin.

DETAILED DESCRIPTION:
The purpose of this protocol is to examine the effects of the sodium-glucose cotransporter 2 (SGLT2) inhibitor canagliflozin on intrarenal transcripts of energy metabolism in adults with type 2 diabetes and early diabetic kidney disease (DKD) via an open-label non-randomized mechanistic trial. This trial will enroll 40 participants who will receive 100 mg of canagliflozin daily for six (6) months in addition to standard of care. The primary objective of this study is to determine whether canagliflozin affects intrarenal transcripts of energy metabolism in adults with type 2 diabetes and early DKD. The primary outcomes measure will be change in transcripts as assessed by single-cell RNA sequencing of kidney biopsy specimens obtained at study entry and after 6 months of study drug. Secondary outcomes include assessing the effects of canagliflozin on structural progression of DKD assessed by morphometric examination of kidney tissue specimens from the paired research biopsies. Additional secondary outcomes include measures of glomerular filtration rate (GFR) and renal plasma flow (RPF) as well as multiparametric kidney MRI. Magnetic resonance imaging of the kidneys will be performed prior to each biopsy to correlate the molecular and structural damage seen at kidney biopsy with the level of perfusion, oxygen availability and fibrosis detected by imaging. Imaging of the kidneys will be done as near to the time of each kidney biopsy as possible. Participants will be followed annually after completion of the mechanistic clinical trial until death or development of end-stage kidney disease.

Of note, participants will be offered the option of staying on the SGLT2 inhibitor free of charge until Jan 2028 to obtain the long-term impact of SGLT2 on GFR and proteinuria. This expansion will be optional and include annual remote visits and extraction of serum creatinine and urine albumin-to-creatinine ratio from their electronic health records.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years. The lower age limit was set so renal function test results would not reflect changes associated with growth.
* Diagnosis of type 2 diabetes for ≥ 3 years.
* Estimated GFR >45 and < 90 ml/min/1.73m2 as determined from the CKD-EPI equation using serum creatinine (Levey et al., 2009).
* A screening urinary albumin-to-creatinine ratio <3000 mg/g.
* Willingness to participate after receiving a thorough explanation of the study.
* Participants receiving a RAAS inhibitor must have been receiving the drug at maximum tolerable dose for at least 3 months prior to the study baseline examination.
* Participants receiving a GLP-1 receptor agonist must have been receiving the drug for at least 3 months prior to the study baseline examination.

Exclusion Criteria:

* Clinically significant disorders of the liver [cirrhosis, portal hypertension, hepatitis, increased bilirubin (≥1.5 mg/dl), active or uncontrolled cardiovascular disease, symptomatic peripheral vascular disease, (i.e. intermittent claudication), pulmonary diseases (including uncontrolled asthma and restrictive or obstructive lung disease requiring therapy), renal-urinary disorders (calculi, urinary tract obstruction, glomerulonephritis, chronic infection), gastrointestinal disorders (nausea, vomiting, diarrhea or anorexia sufficient to cause weight loss or wasting), or hematocrit levels ≤30 percent in women or ≤35 percent in men.
* Prior treatment with SGLT2 inhibitors and unable to perform a wash-out.
* Renovascular or malignant hypertension; uncontrolled hypertension (systolic blood pressure ≥150 or diastolic ≥90 mm Hg)
* Hematuria of unknown etiology. Prior to entry into the study, any participant with hematuria should be evaluated, the etiology established and documented, and treatment rendered as appropriate.
* Chronic debilitating disorders with or without treatment (e.g., systemic lupus erythematosus [SLE], cancer, amyloidosis, and chronic infection) that would interfere with the assessment of kidney function or that might reduce the chances of survival for a sufficient length of time to evaluate the efficacy of treatment.
* Currently receiving a drug regimen that includes steroids, immunosuppressants, or investigational new drugs not associated with this trial.
* Pregnancy. SGLT2 inhibitors are not recommended during the second or third trimester of pregnancy. Moreover, we do not wish to expose pregnant women to conscious sedation that is used during the kidney biopsies or to the intravenous filtration markers iohexol and p-aminohippurate needed for the renal clearance studies. Women of childbearing potential must have a negative pregnancy test prior to entry and every 2 months during the study and agree to using an effective form of contraception throughout the study, such as the oral contraceptive pill or an intrauterine device. Women who are planning a pregnancy in the next three years will be excluded.
* Known hypersensitivity to canagliflozin or iodine.
* Bleeding disorders or requirements for anticoagulation or platelet inhibitors which cannot be safely interrupted, since kidney biopsies cannot be performed safely in these individuals.
* Massive obesity with body mass index ≥45 kg/m². Kidney biopsies are more technically difficult with massive obesity.
* Allergy to iodine-containing contrast material or shellfish.
* Non-diabetic kidney disease - based on clinical history or kidney biopsy examination.
* History of osteoporotic fracture.
* Conditions likely to interfere with informed consent or compliance with the protocol.
* Single kidney; any condition with a single kidney
* Kidney cortex <1 cm (both kidneys)
* Kidney length <8 cm (both kidneys)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Glomerular basement membrane (GBM) width and mesangial expansion | 6 months
  measured by morphometric examination of kidney tissue
Kidney Transcript Changes | 6 months
  Molecular changes measured by change in transcripts as assessed by single-cell RNA sequencing of kidney biopsy specimens

SECONDARY OUTCOMES:
Cortical R2 | 6 months
  Measured by Blood Oxygen Level Dependent (BOLD) MRI; Participants will be scanned in a supine position with a 3T MRI scanner. Spine array and body array receiver coils will be used to maximize image uniformity. Following initial localizer scans, coronal Sec T2-weighted MR images will be obtained to delineate cortical kidney regions. The image acquisition will be respiratory-gated to ensure accurate image co-registration with the respiratory-gated diffusion acquisitions.
Medullary R2 | 6 months
  Measured by Blood Oxygen Level Dependent (BOLD) MRI; Participants will be scanned in a supine position with a 3T MRI scanner. Spine array and body array receiver coils will be used to maximize image uniformity. Following initial localizer scans, coronal Sec T2-weighted MR images will be obtained to delineate medullary kidney regions. The image acquisition will be respiratory-gated to ensure accurate image co-registration with the respiratory-gated diffusion acquisitions.
Renal Perfusion | 6 months
  Measured by Arterial Spin Labeling (ASL)
Glomerular Filtration Rate (GFR) | 3 Hours
  Measured by iohexol clearance; An intravenous (IV) line will be placed, and participants will be asked to empty their bladders. Spot plasma and urine samples will be collected prior to iohexol infusion. Iohexol will be administered through bolus IV injection (36 mg/kg/dose), followed by infusion (15mg/min over 180 min.) An equilibration period of 120 min was used and blood collections for iohexol plasma disappearance were drawn at +120, +150, +180 min.
Renal Plasma Flow (RPF) | 2.5 Hours
  Measured by para-aminohippurate (PAH) clearance; An intravenous (IV) line will be placed, and participants will be asked to empty their bladders. Spot plasma and urine samples will be collected prior to PAH infusion. PAH (2 g/10 mL, prepared by Basic Pharma, with a dose of (16 mg/kg or 12 mg/kg depending on eGFR) will be given slowly over 5 min followed by a continuous infusion of 8 mL of PAH and 42 mL of normal saline at a rate or 7.2 mg/kg/ hr or 5.0 mg/kg/hr for 2 h, depending on eGFR. After an equilibration period, blood will be drawn at 90, 120, and 150 min, and RPF will be calculated as PAH clearance divided by the estimated extraction ratio of PAH, which varies by the level of GFR.

CONTACTS AND LOCATIONS:
Overall Officials: Petter Bjornstad, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No